CLINICAL TRIAL: NCT00713050
Title: Neurophysiological Measurement in Aphasia Treatment
Brief Title: Speech and Language Therapy After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol expired; PI retired
Sponsor: University of Chicago (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Shirley Ryan AbilityLab (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 13785A; 5R01DC007488-05 (NIH)
Record Dates: First submitted 2008-07-09; First posted 2008-07-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Ischemic Stroke
Keywords: stroke; aphasia; imitation; mirror neuron
MeSH Terms: conditions — Ischemic Stroke; Stroke; Aphasia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental (Experimental): Computer-based Aphasia therapy
  Interventions: Behavioral: Imitate Therapy
- Control (Active Comparator): Control Arm - Healthy subjects.
  Interventions: Behavioral: Imitate Therapy

INTERVENTIONS:
Behavioral: Imitate Therapy — Imitation-based computer therapy
  Other Names: Imitate

SUMMARY:
Our overall goal is to advance the state of functional brain imaging in aphasia, and then to apply the method to an intensive, imitation-based treatment for non-fluent aphasia.

DETAILED DESCRIPTION:
Detailed information will follow in the next progress report.

ELIGIBILITY:
Inclusion Criteria:

1. Single ischemic infarction in the MCA territory involving the cerebral cortex (confirmed by CT or MRI)
2. Aphasia
3. Visual attention and language comprehension sufficient to perform imitation fMRI tasks
4. Right handed (prior to stroke)

Exclusion Criteria:

Exclusions to the study are people with cardiac pacemakers, claustrophobia, neurosurgical clips, or cognitive impairments too severe to permit cooperation with cognitive tasks in an MRI scanner.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Changes in scores on Western Aphasia Battery | Four months

CONTACTS AND LOCATIONS:
Overall Officials: Steven Small, M.D., Ph.D., Principal Investigator — University of Chicago
Locations (2):
- United States (2):
  - Solodkin/Small Brain Circuits Laboratory, Irvine, California
  - University of California Irvine, Irvine, California

REFERENCES:
- [Derived] Duncan ES, Schmah T, Small SL. Performance Variability as a Predictor of Response to Aphasia Treatment. Neurorehabil Neural Repair. 2016 Oct;30(9):876-82. doi: 10.1177/1545968316642522. Epub 2016 Apr 6. PMID 27053642